CLINICAL TRIAL: NCT01329406
Title: A Double-Blind, Placebo-Controlled, Enriched Enrollment Randomized Withdrawal Study to Evaluate the Efficacy of Milnacipran in the Treatment of Pain Due to Osteoarthritis
Brief Title: Study to Evaluate the Efficacy of Milnacipran in the Treatment of Pain Due to Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Analgesic Solutions (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Stephen Wright, M.D., Principal Investigator, Analgesic Solutions
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRX001-2010
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis (OA); Milnacipran; Serotonin-norepinephrine reuptake inhibitor (SNRI); Knee pain
MeSH Terms: conditions — Osteoarthritis | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Milnacipran (Experimental): If subjects meet the criteria to enter the Double-Blind Period, they will be randomized at a 1:1 ratio to take either milnacipran or placebo for 4 weeks. The milnacipran arm will take milnacipran at 200mg/day (100mg twice daily).
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator): If subjects meet the criteria to enter the Double-Blind Period, they will be randomized at a 1:1 ratio to take either milnacipran or placebo for 4 weeks. The placebo group will take 1 tablet twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — 1 tablet (100mg) by mouth twice daily for 28 days
  Arms: Milnacipran
Drug: Placebo — 1 tablet by mouth twice daily for 28 days
  Arms: Placebo

SUMMARY:
The present study will aim to evaluate the efficacy of milnacipran in the treatment of pain due to osteoarthritis (OA), that is, to determine whether milnacipran provides superior efficacy to placebo in patients with OA. Milnacipran is a serotonin-norepinephrine reuptake inhibitor (SNRI) that is currently approved in the United States in the treatment of major depressive disorder and fibromyalgia. There is increased evidence to suggest that SNRIs may be effective in the treatment of chronic pain conditions, such as OA.

The hypothesis in this study is that the survival time (time from randomization to loss of efficacy) of milnacipran group is superior to that of placebo group.

DETAILED DESCRIPTION:
The study design is a Double-Blind, Placebo-Controlled, Enriched Enrollment Randomized Withdrawal Study. This means that, upon entry into the study, all subjects will enter an open-label period during which they will take milnacipran for 4 weeks. Subjects will taper their dose up to one 100mg tablet twice daily for a total of 200mg per day. After 4 weeks, the subject will return to the clinic and be re-evaluated.

Only subjects who meet certain criteria are then randomized to continue in the double-blind period of the study. Once a subject is randomized, he or she will take either milnacipran or placebo for another 4 weeks. Following the double-blind period, subjects will be tapered off the study medication and will receive a phone call once each week for 2 weeks for follow-up assessments.

Throughout the study, subjects will complete various questionnaires and other test procedures aimed at sub-typing subjects based on pain mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Be 21-75 years of age and in good general medical and psychological health
* Be able to speak, read, write, and understand English, understand the consent form, complete study related procedures, and communicate with the study staff
* Have a negative urine pregnancy test at screening, and use appropriate birth control
* Have documented painful Osteoarthritis (OA) of at least one knee for at least 6 months; OA should be of Class I-III and meet the American College of Rheumatology (ACR) clinical classification criteria, defined as:

  1. Knee pain and at least 3 of the following 6:

     * Age > 50
     * Morning stiffness < 30 minutes
     * Crepitus on active motion
     * Bony tenderness
     * Bony enlargement
     * No palpable warmth of synovium
  2. The target joint must not contain any type of orthopedic and/or prosthetic device
* Have a target joint pain average of 5 days per week and have an average pain intensity of at least 4/10 on the 0-10 NRS over the last 24 hours prior to screening
* Have stable treatment modalities, e.g. acupuncture, physical therapy
* Be willing to stop taking Non-steroidal Anti-inflammatory drugs (NSAIDs) and opioids for the duration of the study

Exclusion Criteria:

* Are allergic or intolerant to SNRI; have a previous poor response to a SNRI for OA pain; are currently taking an SNRI or tricyclic antidepressant
* Have a body mass index (BMI) >40 kg/m2
* Have an Hospital Anxiety and Depression Scale (HADS) score >12 on either subscale or has an established history of major depressive disorder not controlled with medication
* Have significant pain outside the target knee, including significant hip or back pain. (Bilateral knee OA allowed.)
* Have pain affecting the target knee that is due to any other etiology than OA
* Have documented history of inflammatory arthritis including rheumatoid arthritis
* Have had local injections in target joint within the past 3 months prior to screening
* Have had oral or intramuscular corticosteroids within the past 30 days
* Have had worker's compensation claim, disability, or litigation
* Have a known history of uncontrolled narrow-angle glaucoma
* Have a known history of suicidal ideation
* Use monoamine oxidase inhibitors (MAOI) concomitantly
* Are allergic or intolerant to acetaminophen
* Using opioids 4 or more days per week during the month preceding the screening visit
* Have significant history or renal impairment/failure.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-02 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Time to loss of efficacy in the Double-Blind Period | 28 days
  The time to pain worsening by 30% compared to the value at baseline and a pain score of at least 4 on the 0-10 numerical rating scale on weekly pain assessment. Subjects who drop out due to "lack of efficacy" will be counted as efficacy failures regardless of their pain scores.

SECONDARY OUTCOMES:
Mean change in pain intensity | 28 days
  Mean change in pain intensity on the 0-10 numerical rating scale from baseline in the Double-Blind Period.
Mean change in Western Ontario and McMaster Osteoarthritis Index (WOMAC) scores | 28 days
  Mean change in Western Ontario and McMaster Osteoarthritis Index (WOMAC) scores from Baseline in the Open-Label Period and Double-Blind Period.
The efficacy of milnacipran vs. placebo by time to dropout for all causes | 70 days
The efficacy of milnacipran in the Open-Label Period | 28 days
  The efficacy of milnacipran in the Open-Label Period defined by the change in pain intensity from Baseline to the end of the period and responder proportion.
The difference between milnacipran and placebo in responder proportion in the Double-Blind Period | 28 days
The predictive value of "OA sensory sub-type" for predicting the response to milnacipran vs. placebo | 70 days
Safety and tolerability by monitoring adverse events | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L. Wright, M.D., Principal Investigator — Analgesic Solutions
Locations (1):
- Analgesic Solutions, Natick, Massachusetts, United States